CLINICAL TRIAL: NCT01328639
Title: TeamCare PCN: Collaborative Care for Patients With Diabetes and Depression in Primary Care Networks
Brief Title: TeamCare PCN: Collaborative Care for Diabetes and Depression
Acronym: TeamCare-PCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alliance for Canadian Health Outcomes Research in Diabetes (Other)
Collaborators: Alberta Health & Wellness (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Jeffrey Johnson, Professor, The Alliance for Canadian Health Outcomes Research in Diabetes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Achord 1101-10
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Depression; Depressive Symptoms; Type 2 Diabetes
Keywords: Collaborative care; Diabetes management; Depression management; Primary care
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Participants in this arm will be actively screened for depression and will receive the usual standard care for diabetes from their family physicians based on available clinical practice guidelines.
  Interventions: Other: Usual diabetes and depression care
- TeamCare Depression Intervention (Experimental): Participants in this arm will be actively screened for depression, and will receive care for depression and diabetes based on the collaborative teamcare model for the management of diabetes and co-morbid depression.
  Interventions: Other: TeamCare Depression Intervention

INTERVENTIONS:
Other: TeamCare Depression Intervention — The TeamCare-PCN intervention involves a registered nurse Care Manager (CM), who coordinates collaborative team management for patients with diabetes and depression. The goal of the intervention is to reduce depressive symptoms, achieve targets for cardio-metabolic measures and improve lifestyle behaviours. The intervention includes three phases: (1) managing depression and improving depressive symptoms, (2) managing diabetes and controlling blood glucose, blood pressure and cholesterol, and (3) improving lifestyle behaviours such as healthy eating, physical activity and smoking cessation.
  Other Names: TEAMcare
  Arms: TeamCare Depression Intervention
Other: Usual diabetes and depression care — Usual care of diabetes and depression involves providing care by the family physician based on usual standards of care and available clinical practice guidelines. Usual care does not involve additional active support from the Care Manager.
  Arms: Usual Care

SUMMARY:
Background & Objective: Type 2 diabetes is a complex disease characterized by multiple comorbidities. Depression is one of the most common comorbidities in individuals with diabetes with prevalence rates reaching 30%. Depression complicates diabetes treatment, portends worse outcomes and increases health care costs. One novel approach to managing diabetes with co-morbid depression is a collaborative primary care model involving a multidisciplinary health care team guiding patient-centered care. This model has been tested in the US and showed a significant reduction of depressive symptoms, improved diabetes care and patient-reported outcomes, and saved money. Our aim is to evaluate the implementation of this collaborative care model for type 2 diabetes and comorbid depression within the non-metro Primary Care Network (PCN) setting in Canada.

Intervention: The intervention involves three phases: (1) improving depressive symptoms, (2) improving blood sugar, blood pressure and cholesterol, and (3) improving lifestyle behaviours. The intervention is administered by a CM in collaboration with family physicians, psychiatrists, and internists.

Hypotheses: The TeamCare-PCN intervention will reduce depressive symptoms, achieve targets for cardio-metabolic measures and improve lifestyle behaviours. Furthermore, the investigators anticipate this intervention will be acceptable and implemented in a cost-effective manner in the PCN environment.

Methods: The investigators will employ a mixed-methods approach to our evaluation, using a controlled "on-off" trial design. Our primary analysis will be based on a multivariable scaled marginal model for the combined outcome of depressive symptoms and medical care. Secondary analyses will assess changes in lifestyle behaviours and patient-reported outcomes.

Significance: Our work will serve as a platform upon which an emerging model of primary care can incorporate an effective and cost-effective depression intervention into the management of individuals with type 2 diabetes, and as a framework for implementing and evaluating similar interventions in individuals with other chronic conditions.

DETAILED DESCRIPTION:
I. Brief Overview The over-arching objectives of this study are to implement and evaluate an evidence-based intervention called TeamCare-PCN for individuals with type-2 diabetes and comorbid depression within primary care networks (PCNs). TeamCare-PCN is based on a proven efficacious and cost-saving collaborative primary care model (Katon et al., 2010) which involves a Care Manager (CM) providing active patient management under the supervision of a family physician and consulting psychiatrists and internists. The goal of the intervention is to achieve remission of depression, reach targets for cardio-metabolic measures, and improve lifestyle behaviours.

II. Hypothesis The investigators hypothesize that the TeamCare-PCN intervention will reduce depressive symptoms, achieve targets for cardio-metabolic measures and improve lifestyle behaviours.

III. Setting, Participants, and Sample Size TeamCare-PCN will be conducted in collaboration with 4 PCNs in non-metro Alberta: St. Albert Sturgeon PCN, Leduc/Beaumont/ Devon PCN, Camrose PCN, and Heartland PCN.

We estimate that a minimum total sample size of 120, with 60 in each arm, would provide power of 0.80 to detest a mean difference of 5 points in the PHQ-9, assuming a repeated measures correlation of 0.6, and 2-tailed alpha of 0.05. This sample size also provides more than 80% power (two sided alpha = 0.05) to detect any between-group absolute difference in proportions of 15% or more (e.g., 45% of usual care patients achieve depression remission vs 60% of intervention patients) (Katon et al., 2010). Anticipating a 40% attrition rate, we planned to recruit 168 patients in total across our 4 PCN sites.

IV. Participant Recruitment and Allocation Recruiting participants into TeamCare-PCN involves four steps. i) A screening survey accompanied with an endorsement letter from the PCN and a general information letter. Included in the screen is the PHQ-9.

ii) After potential participants have completed the screening survey and mailed it back to the PCN, staff at the PCN will identify the respondents who are eligible to participate TeamCare-PCN through the responses on the screening survey and by scoring the PHQ-9.

iii) PCN staff will contact eligible participants through a brief phone interview to confirm all eligibility criteria and schedule an initial assessment visit with the CM at the PCN.

iv) CM will meet with the participant, and during the initial assessment, the CM will explain the intervention, provide an intervention-specific information letter and obtain a signed written informed consent from the patient to participate in the study.

Participants will be allocated to study groups using an 'on-off' allocation method. Eligible and consenting respondents who book for an initial assessment with the CM during month 1 will be allocated to the intervention arm (On-group). Those who book the initial assessment in month 2 will be allocated to the usual care arm (Off-group). This allocation process will continue until the target sample size is recruited.

V. Team Care Depression Intervention for Diabetes

A. Patient Management:

Patients entering the intervention will have an initial one-hour appointment with the CM. This first visit will include a bio-psychosocial semi-structured assessment (reviewing medical history, previous treatments for depression and diabetes), patient education, potential treatment options (anti-depressant medications and/or psychotherapy) and developing an overall individualized care plan. The intervention will consist of 3 phases; the first focusing on depression management, the second on cardio-metabolic diabetes management, and the third on general lifestyle modifications. The CM will also have weekly meetings with the consulting specialists to review new cases and patient progress, and then make treatment recommendations to the primary care physician.

B. Training of Care Managers and Specialists:

The CMs and consulting specialists have already received a 2-day training course on the TeamCare-PCN intervention, including the pharmacotherapy of depression and an introduction to psychotherapeutic techniques (i.e. problem solving, behavioural activation, and motivational interviewing), as well as team interactions, roles and responsibilities. An overview of cardio-metabolic diabetes management, including, glucose control, insulin management, blood pressure management and treatment of high lipid levels based on the developed algorithms, was also provided at the training session. TeamCare-PCN training manuals were developed and used in the training sessions, and retained by the CM.

VI. Usual Care All participants in TeamCare-PCN will be actively screened for depression and those allotted to usual care will be identified as such to their family physician. For depression management, patients will receive care from their family physician, without additional active support from the Care Manager.

VII. Data Analysis As the initial focus of the intervention is on the management of depressive symptoms, we have considered the PHQ-9 as a main primary outcome, and will assess changes in PHQ-9 scores over 12-months between groups, adjusting for baseline PHQ-9 score, using a mixed effects multivariate model. For our second primary outcome of improvements in global disease control, we will employ a multivariate model that jointly tests the changes in multiple clinical outcomes, namely A1c, LDL cholesterol and systolic blood pressure. Using the same analytic approach as in the recently published RCT of this intervention, we will apply a scaled marginal model (Katon et al., 2010) to simultaneously compare the change in these continuous outcomes at 12 months, adjusting for the baseline status for each variable. In either primary outcome analyses, the models will be estimated iteratively and the potential correlations among and between outcomes within individuals will be handled using generalized-estimating equation (GEE) models for each outcome.

For all analyses the investigators will employ an intention-to-treat framework for our primary analysis, using a last-observation-carried-forward method of imputation for subjects who do not have complete follow-up data for primary or secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have family physician-identified type 2 diabetes
* 18 years of age or older
* Score >=10 on the PHQ-9
* Speak English and have adequate hearing to complete phone interviews
* Be willing and able to provide written informed consent to participate

Exclusion Criteria:

* Severe and/or terminal physical illness
* Serious and/or severe mental or psychiatric illness
* Pregnant or breastfeeding
* Live in long term care facility
* Already participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 items (PHQ-9) score | Baseline, 3-month, 6-month, 9-month, 12-month
  A remission of depression symptoms is indicated with a PHQ-9 score <10 for a period of three consecutive months.

SECONDARY OUTCOMES:
Change in HbA1c level | baseline, 6-month, 12-month
  Improvement is defined as 10% improvement over baseline
Change in total cholesterol level | baseline, 6-month, 12-month
  Improvement is defined as 10% improvement over baseline
Change in Systolic blood pressure measurement | baseline, 6-month, 12-month
  Improvement is defined as 10% improvement over baseline
Change in self-reported Health Related Quality of Life | Baseline, 6-month, 12-month
  Measured by SF-12-V2 and EQ-5D-5L
Change in Diabetes-specific stress | Baseline, 6-month, 12-month
  Measured by Problem Areas In Diabetes 5-level questionnaire (PAID-5)
Change in Health behaviours | Baseline, 6-month, 12-month
  Includes assessment of smoking behaviours, alcohol consumption, substance use, and physical activity
Change in Self-care management activities | Baseline, 6-month, 12-month
  Measured using the Summary of Diabetes Self Care Activities questionnaire (SDSCA)
Change in Satisfaction with care | Baseline, 12-month
  Measured using the Consumer Assessment of Healthcare Providers and Systems questionnaire (CAHPS), Adult Primary Care 1.0, and the Patient Assessment of Chronic Illness Care questionnaire (PACIC)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Johnson, PhD, Principal Investigator — University of Alberta; Sumit Majumdar, MD, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - Camrose PCN, Edmonton, Alberta
  - Leduc/Beaumont/ Devon PCN, Edmonton, Alberta
  - St. Albert & Sturgeon PCN, Edmonton, Alberta
  - Heartland PCN, Ft Saskatchewan, Alberta

REFERENCES:
- [Background] Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Ludman EJ, Young B, Peterson D, Rutter CM, McGregor M, McCulloch D. Collaborative care for patients with depression and chronic illnesses. N Engl J Med. 2010 Dec 30;363(27):2611-20. doi: 10.1056/NEJMoa1003955. PMID 21190455
- [Background] Jung SH, Ahn C. Sample size estimation for GEE method for comparing slopes in repeated measurements data. Stat Med. 2003 Apr 30;22(8):1305-15. doi: 10.1002/sim.1384. PMID 12687656
- [Background] Majumdar SR, Rowe BH, Folk D, Johnson JA, Holroyd BH, Morrish DW, Maksymowych WP, Steiner IP, Harley CH, Wirzba BJ, Hanley DA, Blitz S, Russell AS. A controlled trial to increase detection and treatment of osteoporosis in older patients with a wrist fracture. Ann Intern Med. 2004 Sep 7;141(5):366-73. doi: 10.7326/0003-4819-141-5-200409070-00011. PMID 15353428
- [Background] Rucker D, Rowe BH, Johnson JA, Steiner IP, Russell AS, Hanley DA, Maksymowych WP, Holroyd BR, Harley CH, Morrish DW, Wirzba BJ, Majumdar SR. Educational intervention to reduce falls and fear of falling in patients after fragility fracture: results of a controlled pilot study. Prev Med. 2006 Apr;42(4):316-9. doi: 10.1016/j.ypmed.2006.01.008. Epub 2006 Feb 20. PMID 16488469
- [Background] Weingarten SR, Riedinger MS, Conner L, Lee TH, Hoffman I, Johnson B, Ellrodt AG. Practice guidelines and reminders to reduce duration of hospital stay for patients with chest pain. An interventional trial. Ann Intern Med. 1994 Feb 15;120(4):257-63. doi: 10.7326/0003-4819-120-4-199402150-00001. PMID 8291818
- [Background] Bell AC, D'Zurilla TJ. Problem-solving therapy for depression: a meta-analysis. Clin Psychol Rev. 2009 Jun;29(4):348-53. doi: 10.1016/j.cpr.2009.02.003. Epub 2009 Feb 26. PMID 19299058
- [Background] Arean P, Hegel M, Vannoy S, Fan MY, Unuzter J. Effectiveness of problem-solving therapy for older, primary care patients with depression: results from the IMPACT project. Gerontologist. 2008 Jun;48(3):311-23. doi: 10.1093/geront/48.3.311. PMID 18591356
- [Background] Mynors-Wallis LM, Gath DH, Lloyd-Thomas AR, Tomlinson D. Randomised controlled trial comparing problem solving treatment with amitriptyline and placebo for major depression in primary care. BMJ. 1995 Feb 18;310(6977):441-5. doi: 10.1136/bmj.310.6977.441. PMID 7873952
- [Background] Cuijpers P, van Straten A, Warmerdam L. Problem solving therapies for depression: a meta-analysis. Eur Psychiatry. 2007 Jan;22(1):9-15. doi: 10.1016/j.eurpsy.2006.11.001. Epub 2006 Dec 27. PMID 17194572
- [Background] Gortner ET, Gollan JK, Dobson KS, Jacobson NS. Cognitive-behavioral treatment for depression: relapse prevention. J Consult Clin Psychol. 1998 Apr;66(2):377-84. doi: 10.1037//0022-006x.66.2.377. PMID 9583341
- [Background] Jacobson NS, Dobson KS, Truax PA, Addis ME, Koerner K, Gollan JK, Gortner E, Prince SE. A component analysis of cognitive-behavioral treatment for depression. J Consult Clin Psychol. 1996 Apr;64(2):295-304. doi: 10.1037//0022-006x.64.2.295. PMID 8871414
- [Background] Jacobson NS, Gortner ET. Can depression be de-medicalized in the 21st century: scientific revolutions, counter-revolutions and the magnetic field of normal science. Behav Res Ther. 2000 Feb;38(2):103-17. doi: 10.1016/s0005-7967(99)00029-7. PMID 10660997
- [Background] Rollnick S, Miller W. What is motivational interviewing? Behavioral Cognitive Psychotherapy 23: 325, 1995.
- [Background] Jacobson N, Martell C, Dimidjian S. Behavioral activation treatment for depression: Returning to contextual roots. Clinical Psychology: Science and Practice 8:255, 2001.
- [Background] Burke BL, Arkowitz H, Menchola M. The efficacy of motivational interviewing: a meta-analysis of controlled clinical trials. J Consult Clin Psychol. 2003 Oct;71(5):843-61. doi: 10.1037/0022-006X.71.5.843. PMID 14516234
- [Background] Butterworth S, Linden A, McClay W, Leo MC. Effect of motivational interviewing-based health coaching on employees' physical and mental health status. J Occup Health Psychol. 2006 Oct;11(4):358-65. doi: 10.1037/1076-8998.11.4.358. PMID 17059299
- [Background] Rubak S, Sandbaek A, Lauritzen T, Christensen B. Motivational interviewing: a systematic review and meta-analysis. Br J Gen Pract. 2005 Apr;55(513):305-12. PMID 15826439
- [Background] Roy J, Lin X, Ryan LM. Scaled marginal models for multiple continuous outcomes. Biostatistics. 2003 Jul;4(3):371-83. doi: 10.1093/biostatistics/4.3.371. PMID 12925505
- [Background] Majumdar SR, Guirguis LM, Toth EL, Lewanczuk RZ, Lee TK, Johnson JA. Controlled trial of a multifaceted intervention for improving quality of care for rural patients with type 2 diabetes. Diabetes Care. 2003 Nov;26(11):3061-6. doi: 10.2337/diacare.26.11.3061. PMID 14578240
- [Background] Majumdar SR, Johnson JA, Bowker SL, Booth GL, Dolovich L, Ghali W, Harris SB, Hux JE, Holbrook A, Lee H, Toth EL, Yale J-F. A Canadian consensus for the standardized evaluation of quality improvement interventions in type 2 diabetes: Development of a Quality Indicator Set. Canadian Journal of Diabetes 29:220-229, 2005
- [Background] Chew LD, Griffin JM, Partin MR, Noorbaloochi S, Grill JP, Snyder A, Bradley KA, Nugent SM, Baines AD, Vanryn M. Validation of screening questions for limited health literacy in a large VA outpatient population. J Gen Intern Med. 2008 May;23(5):561-6. doi: 10.1007/s11606-008-0520-5. Epub 2008 Mar 12. PMID 18335281
- [Derived] Johnson JA, Lier DA, Soprovich A, Al Sayah F, Qiu W, Majumdar SR. Cost-Effectiveness Evaluation of Collaborative Care for Diabetes and Depression in Primary Care. Am J Prev Med. 2016 Jul;51(1):e13-20. doi: 10.1016/j.amepre.2016.01.010. PMID 26947212
- [Derived] Mathe N, Johnson ST, Wozniak LA, Majumdar SR, Johnson JA. Alternation as a form of allocation for quality improvement studies in primary healthcare settings: the on-off study design. Trials. 2015 Aug 25;16:375. doi: 10.1186/s13063-015-0904-x. PMID 26303892
- [Derived] Johnson JA, Al Sayah F, Wozniak L, Rees S, Soprovich A, Qiu W, Chik CL, Chue P, Florence P, Jacquier J, Lysak P, Opgenorth A, Katon W, Majumdar SR. Collaborative care versus screening and follow-up for patients with diabetes and depressive symptoms: results of a primary care-based comparative effectiveness trial. Diabetes Care. 2014 Dec;37(12):3220-6. doi: 10.2337/dc14-1308. Epub 2014 Oct 14. PMID 25315205
- [Derived] Johnson JA, Al Sayah F, Wozniak L, Rees S, Soprovich A, Chik CL, Chue P, Florence P, Jacquier J, Lysak P, Opgenorth A, Katon WJ, Majumdar SR. Controlled trial of a collaborative primary care team model for patients with diabetes and depression: rationale and design for a comprehensive evaluation. BMC Health Serv Res. 2012 Aug 16;12:258. doi: 10.1186/1472-6963-12-258. PMID 22897901